CLINICAL TRIAL: NCT03259243
Title: Port Site Infiltration With Bupivacaine for Reduction of Postoperative Pain in Woman Undergoing Gynecologic Laparoscopy: A Randomized, Factorial, Double-Blind, Controlled Trial
Brief Title: Comparison of Efficacy of Bupivacaine for Relief Postoperative Pain in Women Undergoing Laparoscopic Gynecologic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: RAJLAPGYNE
Record Dates: First submitted 2017-08-19; First posted 2017-08-23 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Pain Score
Keywords: Bupivacaine, Port site infiltration ,Postoperative pain ,Gynecologic laparoscopy
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo group (Placebo Comparator): 0.9%Nacl (Placebo) 10 ml were port site infiltration prior skin incision and prior skin closure Drug: 0.9%Nacl Other Name: NSS
  Interventions: Drug: Bupivacaine Hydrochloride
- Preincision Bupivacaine (Experimental): 0.5% bupivacaine 10 ml (50 mg) were port site infiltration prior skin incision and 0.9%Nacl (Placebo) 10 ml were port site infiltration prior skin closure Drug: 0.5% bupivacaine 10 ml (50 mg) Other Name: Marcaine 0.9%Nacl (Placebo) 10 ml Other Name: NSS
  Interventions: Drug: Bupivacaine Hydrochloride
- Preclosure bupivacaine (Experimental): 0.9%Nacl (Placebo) 10 ml were port site infiltration prior skin incision and 0.5% bupivacaine 10 ml (50 mg) were port site infiltration prior skin closure Other Name: Marcaine
  Interventions: Drug: Bupivacaine Hydrochloride
- Bupivacaine group (Experimental): 0.5% bupivacaine 10 ml (50 mg) were port site infiltration prior skin incision and 0.5% bupivacaine 10 ml (50 mg) were port site infiltration prior skin closure Other Name: Marcaine
  Interventions: Drug: Bupivacaine Hydrochloride

INTERVENTIONS:
Drug: Bupivacaine Hydrochloride — 0.5 Bupivacaine hydrochloride were port site infiltration preincision and preclosure injection
  Other Names: 0.5% Marcaine

SUMMARY:
To comparison of efficacy of Bupivacaine for relief postoperative pain in women undergoing laparoscopic gynecologic surgery

DETAILED DESCRIPTION:
Gynecologic laparoscopic procedures have become more common nowadays because of their benefits in less tissue trauma, less perioperative morbidity and shorter hospital stays compared with laparotomy. But postoperative pain still be the most concerning problems including discomfort at incision sites, Pain due to pneumoperitoneum stretching the intraabdominal cavity and dissection of the abdominal and pelvic viscera.

Visceral pain is at maximal intensity during the first postoperative hours and is exacerbated by coughing, respiratory movements, and mobilization. Because the pain comprises of several factors, multimodal analgesic techniques are needed for effective postoperative analgesia and brought to this study to compare efficacy of Bupivacaine for pain relief postoperatively in women undergoing gynecologic laparoscopic surgery divided into 4 groups including preincision and preclosure Bupivacaine injection collated with placebo group. The result is measurement in postoperative pain score and amount of drug that using to reduce pain

ELIGIBILITY:
Inclusion Criteria:

* Patient who undergoing gynecologic laparoscopic surgery
* Patient who agrees to participate in this study
* Patient able to speak and understand Thai
* Patient able to complete the questionnaire

Exclusion Criteria:

* Patient with history of allergy in any kind anesthetic drug
* Patient who pregnant
* Patient who sign for single port gynecologic laparoscopic surgery or NOTE surgery
* Patient whom the surgery is withhold or canceled
* Patient whom the surgery is converted to laparotomy

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain after surgery | 24-48 hours after surgery
  Postoperative pain score in intervention and placebo groups

SECONDARY OUTCOMES:
Among of pethidine use | within 48 hours
  Among of pethidine use to reduced postoperative pain
Duration of hospital stay | within 7 days
  Duration of hospital stay after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Waetasleem Chema, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No